CLINICAL TRIAL: NCT06163235
Title: Efficacy of a Mobile Application and Semi-attendance Program in Bariatric Surgery: a Randomized Clinical Trial
Brief Title: Efficacy of a Mobile Application and Semi-attendance Program in Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI21/00551
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: Bariatric surgery; Telemedicine; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semi-attendance. (Experimental): This group will follow a semi-attendance program after bariatric surgery.
  Interventions: Other: Obemar platform
- Control group. (No Intervention): This group will follow the conventional controls after bariatric surgery.

INTERVENTIONS:
Other: Obemar platform — Online platform for education and follow-up
  Arms: Semi-attendance.

SUMMARY:
BACKGROUND: Applications for mobile devices in patients with obesity offer a great opportunity to improve the quality of care and the monitoring of patients in bariatric surgery programs. This is especially pressing in the context of an increasing prevalence of obesity, and longer waiting lists in bariatric surgery programs.

OBJECTIVES: The main objective is to evaluate the efficacy of a digital platform on mobile devices in obesity and bariatric surgery programs. Investigators will compare weight loss at 12 months after surgery in patients in the standard of care program and those in a semi-attendance program with digital support through a mobile application. As secondary objectives, it will be compared: (1) the number medical complications, the quality of life and satisfaction, physical activity, diet and attrition at 12 months after surgery. Investigators will also study the patient interaction with the platform and social networks.

TRIAL DESIGN: Randomized, non-inferiority clinical trial with a 12-month follow-up.

METHODS: 72 patients will be randomized (1: 1) to standard of care program and to semi-attendance program with digital support from the bariatric surgery program waiting list. Inclusion criteria: age between 18 and 60 years, body mass index between 35-50kg/m2, candidates for the sleeve gastrectomy technique, and possession of a mobile device. Participants will be evaluated before and 12 months after surgery. Variables: anthropometric measurements, medical complications during follow-up, quality of life, diet and physical activity questionnaires. Primary endpoint: weight loss 12 months after surgery.

DETAILED DESCRIPTION:
Introduction

In Spain, the prevalence of obesity in adults has increased from 14% to 21.6% between 2003 and 2016. The category of obesity that has increased the most is severe obesity. Forecasts for the next ten years maintain that the increase will continue.

The two main problems of current bariatric surgery programs are the saturation of healthcare resources, and the losses to follow-up and long-term treatment adherence. Patients on the waiting list for bariatric surgery and who have completed the preoperative program can be found for a long period in a situation where there is no proactive specialized follow-up and without ability to consult with a multidisciplinary team.

On the other hand, loss to follow-up is another unresolved problem currently in bariatric units. Longer follow-up by specialized units has been associated with greater long-term weight loss. However, the loss to follow-up at 5 years can be as high as 40%, and even higher in the longer term. The already existing saturation of resources prior to the COVID-19 pandemic and the new limitations generated by it, have highlighted the need to reformulate bariatric surgery programs.

In this sense, the incorporation of digital platforms and applications for mobile devices can contribute to the digital transformation of the health care system to severe obesity.

Digitalisation offers numerous possibilities to provide educational material to patients, monitor their physical activity, or a more frequent and personalized follow-up.

The use of mobile applications has proven to be effective in losing weight in overweight patients without severe obesity, and in promoting the practice of physical activity. However, the majority of published studies use commercial mobile applications with very limited functionalities, so it has not been possible to evaluate all the multidisciplinary aspects involving a real bariatric patient follow-up.

To sum up, there is a lack of studies that analyze the full potential of digital platforms in patients with obesity and bariatric surgery. This project wants to design and test a mobile application in a randomized clinical trial, with multiple functionalities for mobile devices and that at the same time provides a safe and effective digital environment for patients included in bariatric surgery programs. Likewise, we want to evaluate the possible usefulness of the digital for the follow-up of these patients.

Methods and analysis Primary objective Assess the non-inferiority of a semi-presential program (40% reduction in face-to-face visits) with digital support compared with the conventional face-to-face follow-up program of the bariatric surgery program in the weight loss at 12 months after bariatric surgery.

Secondary objective

1. To compare postoperative weight loss at 3 and 6 months after bariatric surgery by semi-presential follow-up with digital support versus conventional face-to-face visit program.
2. To compare other secondary efficacy parameters at 12 months in the two follow-up arms:

2.1. Medical-surgical complications after surgery. 2.2. The quality of the diet. 23. The degree of physical activity. 2.4. Quality of life and degree of satisfaction with treatment. 2.5. Follow-up adherence. 2.6. Cost analysis.

Patients and public involvement Neither patients nor the public are involved in the conception, design or conduct of the study.

Study design Non-pharmacological, open-label, single center clinical trial to assess the impact of a semi-presential program with digital support through a mobile application in bariatric surgery programs.

Eligibility criteria for participants Patients suffering from severe obesity, candidates for treatment through bariatric surgery, on the waiting list for surgery at the Hospital del Mar in Barcelona. The inclusion of participants will be performed after obtaining the written informed consent approved by the ethical committee.

A) Inclusion criteria: patients between 18 and 65 years old who accept and understand the characteristics of the semi-presential program with digital support; BMI between 35-50kg/m2; sleeve gastrectomy, Roux-en-Y gastric bypass and SADI-S candidates.

B) Exclusion criteria: non-controlled psychiatric disorder; pregnancy desire in the next 12 months; do not have mobile devices; do not understand Spanish.

Blinding There will be no blinding with regard to the type of follow-up: patients as well as physicians and dietitians assessing follow-up data will be informed of the procedure performed.

Recruitment Participants will be recruited from the BS program at the Hospital del Mar, Barcelona. Patients who meet the NIH criteria for BS (BMI ≥40 kg/m2 or ≥35 kg/m2 with significant obesity-related comorbidities) and who express the desire to undergo BS will be referred to the BS unit from primary care units.

Inclusion visit(?) Preoperative management and postoperative follow-up

Prior to bariatric surgery, different examinations will be performed (abdominal ultrasound, functional respiratory tests and gastroscopy) and results evaluated by a multidisciplinary team including dietitian, surgeon and endocrinologist. Ten days prior to surgery, a very low-calorie diet will be prescribed to achieve additional weight loss.

The control group will make 30 face-to-face visits (16 preoperative and 14 postoperative), while the intervention group will make 11 face-to-face visits, 10 through online support and 9 telematic visits (7 face-to-face visits, 7 through online support and 2 telematic visits during the preoperative period and 4 face-to-face visits, 3 through online support and 7 telematic visits in the postoperative period). This is 40% fewer face-to-face visits in the second group. Both groups will have at their disposal the interaction with the medical team through social networks.

Randomization All patients who meet the inclusion criteria and do not present exclusion criteria will be randomized 1:1 in two parallel arms between the control group (face-to-face) and the intervention group (semi-presential).

Surgical procedures The present study contemplates laparoscopic Roux-en-Y gastric bypass, sleeve gastrectomy and SADI-S.

In order to avoid variability of response depending on the surgical technique and BMI, the study will be restricted to patients with obesity grade II-III (BMI between 35 and 50 kg/m2) who are candidates to bariatric surgery as a non-sequential technique.

The procedures are performed using a laparoscopic approach and involves a hospital stay of 1-2 days. All the procedures will be performed by the same surgical team.

Outcome definition

1. Main variable: weight loss at 12 months after bariatric surgery. It will be determined as the percentage of total weight loss [%TWL= 100 x (Basal weight - Weight 12 months) / Basal weight].
2. Secondary variables:

I. Medical-surgical complications: the variables corresponding to the biochemical and hematological determinations will be collected prior and 12 months after surgery. Surgical complications will be recorded using ordinal variables according to the Clavien-Dindo scale during the first 30 days after surgery. From the 30th day all complications will be recorded as a nominal variable. We will also record non-planned care activity that will include the number of emergency visits, readmissions and reinterventions.

II. Diet quality: it will be recorded using the "Short Diet Quality Screener" (sDQS) questionnaire validated in Spanish, before and 12 months after surgery.

III. Degree of physical activity: it will be evaluated using the reduced version of the physical activity questionnaire of Minnesota (Minnesota Leisure Time Physical Activity Questionnaire) before and 12 months after surgery, validated in Spanish. IV. Degree of satisfaction and quality of life: the first one will be recorded using a categorical scale. The second one Through the SF-36 quality of life questionnaire. V. Loss to follow-up: it will be collected as absence of visits for more than 6 months.

VI. To analyze the costs of both programs we will use the variables that encompass the set of healthcare activities carried out on all the patients attended, both in the emergency room, admissions, surgery and also in the outpatient setting, tests and examinations.

VII. To evaluate the behavior of patients in social networks and the same mobile application, we will use the variables of the length of the messages, the frequency of repetition of words, the periodicity of connection and participation in social networks, as well as the type of semantics used. In this sense, the team has a wide experience in the selection and collection of variables from social networks through the Application Programming Interface (API). The categorization of the digital phenotype according to the combination of variables can help to detect possible patterns of digital behavior that are capable of predicting the evolution of the disease.

Anthropometric parameters BMI will be calculated as weight in kilograms divided by the square of height in meters. Weight loss will be measured as percentage of total weight loss [%TWL= 100 x (Basal weight - Weight 12 months) / Basal weight].

Sample size Sample size has been calculated based on the primary objective to demonstrate the non-inferiority between treatments. Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a unilateral contrast, 36 subjects are required in the first group and 36 in the second to detect a difference equal to or greater than 5 units in the %TWL. The common standard deviation is assumed to be 8. A loss-to-follow-up rate of 10%. As a contingency plan for possible missing values (missing data) in the covariates, we plan to carry out a multiple imputation analysis if necessary.

Data analysis

1. Primary outcome:

   The analysis of weight loss at 12 months will be carried out using a model of multivariate analysis of variance including type of relationship with patients and gender as factors, and age and initial BMI as covariates. Likewise, a multiple linear regression model will be developed with these variables.
2. Secondary objectives will be evaluated respectively by:

   1. Post-surgery complications will be analyzed using Fisher's exact tests.
   2. The quality of the diet will be analyzed by a t-Student for independent samples.
   3. Physical activity levels will be compared with the t-Student test for independent samples and for matched-samples.
   4. The satisfaction and quality of life will be compared with a t-Student for independent samples.
   5. Adherence to follow-up will be evaluated with a Poisson regression.
   6. Economic analysis: Hospital del Mar has a cost information system based on costs (Full-costing) and distribution of costs by activities (ABC), which allows evaluating the set of assistance activities carried out on all the patients attended, both in emergencies, admissions, surgery and also in the outpatient setting, tests and explorations. For any patient selected in the study,

Ethics and dissemination

The study will be conducted in accordance with the basic principles of protection of rights and dignity of the human being, as stated in the Helsinki Declaration and with current regulations. All the information obtained will be treated confidentially in compliance with the personal data protection legislation (Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos Personales y garantía de los derechos digitales). Participants will sign their informed consent to participate in the study. Ethics approval has been granted by the Parc de Salut Mar Ethics Committee (2022-9964-I). The study and its conclusions regarding the primary and secondary objectives will be presented as manuscripts submitted for peer-reviewed journal publication.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 35-50kg/m2
* Bariatric surgery candidates

Exclusion Criteria:

* Non-controlled psychiatric disorder
* Pregnancy desire in the next 12 months
* Do not have mobile devices (smartphone)
* Language barrier with Spanish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year
  The percentage of total weight loss at 12 months after bariatric surgery.

SECONDARY OUTCOMES:
Medical-surgical complications. | 1 year
  The variables corresponding to the biochemical and hematological determinations will be collected prior and 12 months after surgery. Surgical complications will be recorded using ordinal variables according to the Clavien-Dindo scale during the first 30 days after surgery. From the 30th day all complications will be recorded as a nominal variable. We will also record non-planned care activity that will include the number of emergency visits, readmissions and reinterventions.
Diet quality. | 1 year
  It will be recorded using the "Short Diet Quality Screener" (sDQS) questionnaire validated in spanish, before and 12 months after surgery.
  The total possible score ranges from 18 to 54, where higher scores mean worse results.
Degree of physical activity. | 1 year
  It will be evaluated using the reduced version of the physical activity questionnaire of Minnesota (Minnesota Leisure Time Physical Activity Questionnaire) before and 12 months after surgery, validated in spanish. Metabolic equivalent of task (MET) are measured through this questionnaire. More METs means more exercise.
Degree of satisfaction and quality of life. | 1 year
  The first one will be recorded using a categorical scale. The second one Through the Short Form -36 quality of life questionnaire. Score ranges from 0 to 100, meaning 0 the worst result and 100 the best.
Loss to follow-up. | 1 year
  Number of partiticpants who skip visits for more than 6 months.
Cost analysis. | 1 year
  We will use the variables that encompass the set of healthcare activities carried out on all the patients attended, both in the emergency room, admissions, surgery and also in the outpatient setting, tests and examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Casajoana, PhD, Principal Investigator — Hospital del Mar Research Institute

IPD SHARING:
Plan to Share IPD: No